CLINICAL TRIAL: NCT05926752
Title: Photobiomodulation Therapy for Myofascial Pelvic Pain: A Randomized Clinical Study
Brief Title: Photobiomodulation for Myofascial Pelvic Pain
Acronym: PMPP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Orlando VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Mario Castellanos, Physician, Orlando VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1591638
Record Dates: First submitted 2023-06-09; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Pelvic Pain; Levator Ani Syndrome; Spastic Pelvic Floor Syndrome; Chronic Pelvic Pain Syndrome; Myalgia of Pelvic Floor
Keywords: photobiomodulation; pelvic floor physical therapy; chronic pelvic pain; spastic pelvic floor syndrome; levator ani syndrome; myalgia of pelvic floor
MeSH Terms: conditions — Pelvic Pain; Levator syndrome; Vaginismus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Photobiomodulation (Active Comparator): The participant will be treated with intravaginal SoLá photobiomodulation therapy for a total of nine treatments (two treatments a week). Each treatment lasting 5 minutes.
  Interventions: Device: SoLá therapy
- Pelvic Floor Physical therapy (Active Comparator): The participant will be treated with pelvic floor physical therapy once a week for 8 weeks. Physical therapy involves standard approach of manual therapy including trigger point release, soft tissue mobilization, stretching, biofeedback, breathing techniques, relaxation yoga, and therapeutic exercises.
  Interventions: Other: Pelvic floor physical therapy

INTERVENTIONS:
Device: SoLá therapy — SoLá therapy is a photobiomodulation device that works by stimulating mitochondria, soothing tense muscles, and promotes healing.
  Arms: Photobiomodulation
Other: Pelvic floor physical therapy — Physical therapy is manual myofascial release, muscles stretches, and exercises designed to help myofascial pelvic pain
  Arms: Pelvic Floor Physical therapy

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy of photobiomodulation of the pelvic floor muscles in female Veterans with chronic pelvic pain. The main questions it aims to answer are:

* Is there a difference in reduction in overall pelvic pain between women who undergo photobiomodulation compared to women who received pelvic floor physical therapy?
* Is there a difference in compliance with therapy between the two groups? Participants will be randomized to treatment with either 9 treatments of photobiomodulation (two treatments per week) or 8 weeks of pelvic floor physical therapy (one treatment a week). Researchers will compare both groups to see if there is a difference in overall pelvic pain reduction.

DETAILED DESCRIPTION:
Background:

Myofascial pelvic pain (MFPP) is defined as pain in the pelvic floor muscles, the pelvic floor connective tissue, and the surrounding fascia. Standard treatment options of MFPP include pharmacotherapy and pelvic floor physical therapy (PT). In severe cases (approximately 25%) who are not responsive to therapy, pudendal blocks and trigger point injections (TPs) may be used to temporarily alleviate pain and improve function. However, these are more invasive and may require anesthesia. Photobiomodulation therapy (PBMT) delivered by a low-level laser emitter has recently emerged as a treatment option for musculoskeletal disorders such as neck and low back pain. In patients with vaginal musculoskeletal pain, PBMT is also thought to be effective with minimal side-effects. SoLá is low-level pelvic laser emitter / photobiomodulation device that has FDA approval for intravaginal use to specifically treat myofascial pelvic pain and chronic pelvic pain. Although it is FDA approved and thought to be effective and less invasive, photobiomodulation using SoLá has not been rigorously studied in randomized controlled trials (RCTs).

Study Aims:

The primary aim is to evaluate the efficacy of SoLá pelvic therapy by comparing reduction in overall pelvic pain between women who undergo 9 treatments of photobiomodulation with SoLá (approximately 1 treatment twice a week), compared to women who receive standard pelvic floor PT once a week for 8 weeks. The secondary aim is to compare dyspareunia, pain with sitting, and compliance with therapy between the two groups.

Study Design and Methods:

The investigators will conduct a RCT comparing overall pelvic pain (primary outcome), dyspareunia, and pain with sitting in women who receive PBMT with SoLá (group 1) vs. women who receive pelvic floor PT (group 2). Twenty-eight total participants will be randomized to either study group after providing informed consent. After enrollment, participants will be treated with 8 weekly treatments of pelvic PT or 9 treatments of SoLá (administered twice weekly). Patient outcomes will be evaluated at baseline (before treatment 1), midway through their treatment (before treatment 5 of SoLá and treatment 5 of PT), and at the end of their treatment (1-2 weeks after treatment 8 of PT/treatment 9 of SoLá and 3 months after treatment 8 of PT/treatment 9 of SoLá). Pain levels will be assessed using the Short Form McGill Pain Questionnaire (SF-MPQ) which assesses sensory and affective components of pain, Pain Interference Short Form which evaluates the effect of pain on quality of life, and pain severity on a 1-10cm Visual Analog Scale (VAS).

Anticipated Results:

The investigators hypothesize that women who undergo PBMT will demonstrate greater improvements in all pain outcomes when compared to pelvic floor PT.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed MFPP
* Age ≥ 18
* Able to provide informed consent
* English speaking
* Agree not to participate in any other form of treatment of myofascial pelvic pain for 3 months after end of trial

Exclusion Criteria:

* Prior pelvic floor physical therapy or SoLá therapy for pelvic pain
* Pregnancy documented by urine or blood
* Taking drugs that have heat- or light- sensitive contraindications
* Reporting decreased sensation in the vagina or rectum or if they are found to have abnormalities on the external neurosensory exam of the vagina
* Have a known history of cancer of the cervix, vagina, uterus, bladder, or vulva or suspected to have neoplasia or pre-cancerous lesions
* Have an active infection of the bladder, vagina, vulva, or urethra
* Have active vaginal bleeding or blood in the vaginal canal
* Have evidence of active vaginal trauma, ulcerations, erosions, or other evidence of vaginal and vulvar skin breakdown
* Cannot tolerate vaginal examination either due to discomfort, pain or history or traumatic experience

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2021-10-27 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Pelvic Pain Intensity | 3 months post treatment
  Change pelvic pain intensity using a 0-10cm visual analog scale. High score means a worse outcome.

SECONDARY OUTCOMES:
Intensity of Dyspareunia | 3 months post treatment
  Change in dyspareunia intensity using a 0-10cm visual analog scale. High score means a worse outcome.
Intensity of pain with sitting | 3 months post treatment
  Change in intensity of pain with sitting using a 0-10cm visual analog scale. High score means a worse outcome.
Pain interference | 3 months post treatment
  change in the score from the Pain Interference Short Form 8A PROMIS® (Patient-Reported Outcomes Measurement Information System) Health Organizations questionnaire. High score is associated with worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Orlando VA Medical Center, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No
Final data sets underlying publications resulting from the proposed research will not be shared outside VA, except as required under the Freedom of Information Act (FOIA).

REFERENCES:
- [Background] Bonder JH, Chi M, Rispoli L. Myofascial Pelvic Pain and Related Disorders. Phys Med Rehabil Clin N Am. 2017 Aug;28(3):501-515. doi: 10.1016/j.pmr.2017.03.005. PMID 28676361
- [Background] Lamvu G, Carrillo J, Witzeman K, Alappattu M. Musculoskeletal Considerations in Female Patients with Chronic Pelvic Pain. Semin Reprod Med. 2018 Mar;36(2):107-115. doi: 10.1055/s-0038-1676085. Epub 2018 Dec 19. PMID 30566976
- [Background] Cichowski SB, Rogers RG, Komesu Y, Murata E, Qualls C, Murata A, Murata G. A 10-yr Analysis of Chronic Pelvic Pain and Chronic Opioid Therapy in the Women Veteran Population. Mil Med. 2018 Nov 1;183(11-12):e635-e640. doi: 10.1093/milmed/usy114. PMID 29788455
- [Background] Fuentes-Marquez P, Cabrera-Martos I, Valenza MC. Physiotherapy interventions for patients with chronic pelvic pain: A systematic review of the literature. Physiother Theory Pract. 2019 Dec;35(12):1131-1138. doi: 10.1080/09593985.2018.1472687. Epub 2018 May 14. PMID 29757068
- [Background] FitzGerald MP, Payne CK, Lukacz ES, Yang CC, Peters KM, Chai TC, Nickel JC, Hanno PM, Kreder KJ, Burks DA, Mayer R, Kotarinos R, Fortman C, Allen TM, Fraser L, Mason-Cover M, Furey C, Odabachian L, Sanfield A, Chu J, Huestis K, Tata GE, Dugan N, Sheth H, Bewyer K, Anaeme A, Newton K, Featherstone W, Halle-Podell R, Cen L, Landis JR, Propert KJ, Foster HE Jr, Kusek JW, Nyberg LM; Interstitial Cystitis Collaborative Research Network. Randomized multicenter clinical trial of myofascial physical therapy in women with interstitial cystitis/painful bladder syndrome and pelvic floor tenderness. J Urol. 2012 Jun;187(6):2113-8. doi: 10.1016/j.juro.2012.01.123. Epub 2012 Apr 12. PMID 22503015
- [Background] Chow RT, Johnson MI, Lopes-Martins RA, Bjordal JM. Efficacy of low-level laser therapy in the management of neck pain: a systematic review and meta-analysis of randomised placebo or active-treatment controlled trials. Lancet. 2009 Dec 5;374(9705):1897-908. doi: 10.1016/S0140-6736(09)61522-1. Epub 2009 Nov 13. PMID 19913903
- [Background] Glazov G, Yelland M, Emery J. Low-level laser therapy for chronic non-specific low back pain: a meta-analysis of randomised controlled trials. Acupunct Med. 2016 Oct;34(5):328-341. doi: 10.1136/acupmed-2015-011036. Epub 2016 May 20. PMID 27207675
- [Background] Lev-Sagie A, Kopitman A, Brzezinski A. Low-Level Laser Therapy for the Treatment of Provoked Vestibulodynia-A Randomized, Placebo-Controlled Pilot Trial. J Sex Med. 2017 Nov;14(11):1403-1411. doi: 10.1016/j.jsxm.2017.09.004. Epub 2017 Sep 29. PMID 28970071